CLINICAL TRIAL: NCT04437953
Title: Clinical Trial of Avatrombopag for Thrombocytopenia in Cancer, A Phase II Single Arm Study
Brief Title: Avatrombopag for Thrombocytopenia in People With Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Sobi, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-483
Record Dates: First submitted 2020-06-17; First posted 2020-06-18 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Thrombocytopenia; Cancer; Liver Diseases
Keywords: Avatrombopag; 19-483
MeSH Terms: conditions — Thrombocytopenia; Neoplasms; Liver Diseases | interventions — avatrombopag

STUDY DESIGN:
Intervention Model Description: A Phase II single arm study will be an open label study examining the use of Avatrombopag.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Avatrombopag (Experimental): Patients will receive an initial dose of Avatrombopag 60 mg on Day 1.Starting on Day 2, the dose will be Avatrombopag 20 mg daily.
  Interventions: Drug: Avatrombopag

INTERVENTIONS:
Drug: Avatrombopag — Patients will receive an initial dose of Avatrombopag 60 mg on Day 1. Starting on Day 2, the dose will be Avatrombopag 20 mg daily. Once a patient has reached a platelet target of > 100,000/mcL patients can initiate systemic cancer therapy. Avatrombopag will be continued as maintenance (subscript "m") and titrated weekly with a goal to maintain a platelet count of ≥ 100,000/mcL during administration of systemic cancer therapy. Duration of maintenance therapy will be at least 12 weeks (indicated by Week 1m, Week 2m, … 12m) starting from time of platelet correction and resumption of systemic cancer therapy. End of Treatment (EOT) is up to 15 weeks on study Week 12m.

SUMMARY:
This study will test whether avatrombopag is an effective treatment for thrombocytopenia in people who have both cancer and a liver disease (such as cirrhosis, cholangitis, or hepatitis). Researchers will look at whether giving participants avatrombopag for 3 weeks can raise their platelet levels enough for them to begin chemotherapy. The study will also test whether avatrombopag can continue to be effective against thrombocytopenia while participants are on chemotherapy for 12 weeks or longer. In addition, researchers will determine how safe the study drug is in participants.

ELIGIBILITY:
Inclusion Criteria:

* Patients with history of locally advanced or metastatic solid tumor, with a plan to initiate cancer directed systemic therapy for adjuvant or palliative purposes.
* 18 years of age or greater
* Known liver disease attributed to one of the following:

  1. Chronic HBV and/or chronic HCV with Cirrhosis
  2. Alcoholic Cirrhosis
  3. Nonalcoholic Fatty Liver Disease with Cirrhosis
  4. Primary Biliary Cholangitis
  5. Primary Sclerosing Cholangitis
  6. Autoimmune Hepatitis
  7. Hereditary Hemochromatosis
  8. Wilsons Disease
  9. Alpha-1 Antitrypsin Deficiency
  10. Congestive Hepatopathy
  11. Cirrhosis or known pre-existing liver dysfunction of unknown cause, or not otherwise specified
* No specific Child-Pugh Score will be required for eligibility.
* Patients with liver involvement with primary or metastatic cancer are eligible, if the patient also has a diagnosis from list in eligibility
* Platelet count of < 80,000/mcL at time of enrollment, and no platelet count ≥ 80,000/mcL in the 4 weeks prior to enrollment. A platelet count ≥ 80,000/mcL in the prior 4 weeks within 72 hours of a platelet transfusion will not make a patient ineligible.
* No prior cancer directed therapy that is cytotoxic, marrow suppressive, or has thrombocytopenia as a known common side effect in the past 12 months.

  a. For purposes of this study, cytotoxic/marrow suppressive systemic cancer therapy drugs will include: i. Nucleoside Analogue, including gemcitabine and fluorouracil ii. Carboplatin or cisplatin iii. Anthracycline iv. Alkylating agent v. Other cancer directive therapies with thrombocytopenia as a known common toxicity even if not cytotoxic b. If a patient has received cytotoxic systemic cancer therapy at any time in the past, then patients will be evaluated for myelodysplastic syndrome and leukemia prior to enrollment
* ECOG Performance status ≤ 2.

Exclusion Criteria:

* History of immune causes of thrombocytopenia (ITP).
* Presence of leukemia or myelodysplastic syndrome.
* Known bone metastases sufficient to result in at least one site of cortical bone destruction, osteolytic lesions, or osteoblastic lesions, on radiologic imaging.
* Patients who have previously received thrombopoietin mimetics such as romiplostim, eltrombopag, etc.
* Patients who require emergent systemic cancer therapy will be excluded.
* Patients who require emergent radiation therapy will be excluded.

  a. Note: Concomitant radiation therapy with systemic cancer therapy is permitted.
* Pancytopenia at enrollment (Hemoglobin <9 g/dL and/or Absolute Neutrophil Count < 1500/mcL).

  a. G-CSF and Red Blood Cell transfusions to treat anemia and neutropenia and achieve adequate hemoglobin and ANC are permitted.
* Patients with serum sodium ≤130 mEq/L will be excluded.
* Patients with a known bleeding disorder or platelet dysfunction will be excluded

  1. Baseline Prothrombin Time (PT) that is greater than 2" above the upper limit of normal.
  2. Activated Partial Thromboplastin Time (aPTT) that is greater than 3" above the upper limit of normal.
* Patients with known genetic prothrombotic conditions (Factor V Leiden, Prothrombin 20210A, Antithrombin deficiency or Protein C or S deficiency) or history of antiphospholipid syndrome.
* Patients on anticoagulation or NSAIDs within 7 days of enrollment will be excluded, with the exception of celecoxib.
* Patients with concurrent lymphoma will be excluded.
* Patients will be excluded if they have a known pre-existing portal vein thrombus, mesenteric thrombus, or splenic thrombus that is not in the context of tumor invasion. Pre-existing tumor-associated portal vein thrombus, mesenteric thrombus, or splenic thrombus are not excluded.
* Potential drug interactions: Moderate or strong inducers of cytochrome p450 (CYP)2C9 or CYP3A4/5 and use of dual moderate inhibitors of CYP2C9 and CYP3A4/5 may interact with Avatrombopag. Patients will be ineligible if they are receiving any of the following drugs:

  1. Itraconazole, Fluconazole, Rifampin, Cyclosporine, Verapamil
  2. If patients had been previously receiving the above drugs, the last dose must have been administered 7 or more days before initiation of the first dose of Avatrombopag.
* Females who are pregnant or breastfeeding or planning to become pregnant or breastfeed during treatment and for an additional 30 days after treatment discontinuation or longer if required by prescribing information for systemic cancer therapy received during the study will be excluded.
* Patients unwilling to use highly effective contraception during the study period and for the duration required by prescribing information for systemic cancer therapy (ies) administered during the study.

  1. If a woman, before entry she must be: postmenopausal (for at least 12 months), or surgically sterile (have had a total hysterectomy or bilateral oophorectomy, tubal ligation, or otherwise be incapable of pregnancy), or practicing a highly effective method of birth control, if sexually active, including hormonal prescription oral contraceptives,contraceptive injections, contraceptive patch, intrauterine device, double-barrier method for less effective methods of contraception (eg,condoms, diaphragm, cervical cap, or sponge with spermicidal foam, cream, or gel), or male partner sterilization, consistent with local regulations regarding use of birth control methods for subjects participating in clinical trials, for the duration of their participation in the study, or not heterosexually active.

     Note: subjects who are not heterosexually active at screening must agree to utilize a highly effective method of birth control if they become heterosexually active during their participation in the study.
  2. If a man, must agree to use an adequate contraception method as deemed appropriate by the investigator (eg, vasectomy, condoms, partner using effective contraception).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2020-12-03 (Actual)

PRIMARY OUTCOMES:
Number of patients who achieve platelet counts of ≥ 100,000/mcL | within 3 weeks of treatment
  the platelet count is ≥ 100,000/mcL, this will be considered successful achievement of the primary endpoint

SECONDARY OUTCOMES:
Number of patients who can undergo systemic cancer therapy without more than one dose delay or dose reduction | 12 weeks
  without platelets dropping below 100,000/mcL on the day of the start of next scheduled cycle of systemic cancer therapy

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Soff, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm